CLINICAL TRIAL: NCT01539200
Title: Effects of 6-months Once Daily Nutritional Supplementation in Combination With a Once Weekly Jacques-Delacroze Eurhythmics Training (NUDAL) on Functionality, Probability of Independence and/or Functional Reserve Among Community-dwelling Seniors
Brief Title: Effects of Daily Nutritional Supplementation in Combination With a Eurhythmics Training (NUDAL)
Acronym: NUDAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUD1051
Record Dates: First submitted 2012-02-15; First posted 2012-02-27 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Improvement of Functionality

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: JDR
- Oral Nutritional Supplement (ONS) and JDR (Active Comparator)
  Interventions: Dietary Supplement: ONS+JDR

INTERVENTIONS:
Dietary Supplement: ONS+JDR — Oral Nutritional Supplement with Jacques-Delacroze Eurythmic training
  Arms: Oral Nutritional Supplement (ONS) and JDR
Dietary Supplement: JDR — Jacques-Delacroze Eurythmic training with placebo ONS
  Arms: Control

SUMMARY:
Malnutrition and lack of regular exercise are often found in older adults and have been identified as important risk factors for independence loss and nursing home admission in older community-dwelling adults.

Existing evidence suggests that high protein nutritional supplements can increase skeletal muscle protein synthesis following exercise in older individuals. However, increase of muscle strength by resistance training does not decrease the rate of falls and is not necessarily linked to an improvement of physical function. In contrast to resistance training, T'ai Chi, dance and eurhythmics have been shown to decrease fall incidence and improve mobility and physical function in older adults. The investigators will examine the combination of eurhythmics and high protein nutritional supplements.

The aim of the study is to investigate whether there is an increase in normal walking velocity due to the nutritional supplement on top of once weekly Jacques-Delacroze Eurhythmics training.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling males and females, aged ≥ 65 years
* Able to walk unassisted for 15 meters
* MMSE ≥ 24 points
* Having obtained his/her informed consent

Exclusion Criteria:

* Serum 25(OH) Vitamin D > 100 nmol/L from the blood sampling at Screening
* Current regular (defined as >3x /week) use of high protein oral nutritional supplements
* Milk protein allergy (Lactose intolerance)
* Severe visual impairment (corrected near vision <0.2 in both eyes)
* Severe neurological, orthopaedic, rheumatologic or psychiatric illness causing inability to understand or follow task instructions or to walk 15 meters without assistance (if clinically questionable, final decision will be made by a senior physician)
* Terminal illness with life expectancy less than 12 months, as determined by a physician

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Normal walking velocity | 6 months
  The primary objective is to demonstrate in older adults receiving a once weekly Jacques-Delacroze Eurhythmics (JDR) training for six months, that a once daily nutritional supplementation increases normal walking velocity compared with placebo. The primary endpoint of this study is normal walking velocity (NW velocity, in cm/s) six months after the onset of the treatment.

SECONDARY OUTCOMES:
Quality of Life and Nutritional status | baseline, 3 months, 6 months
  The secondary objectives of the research project are to compare the effects of the NUDAL intervention versus JDR alone, on changes in functional measures, nutritional status and health-related quality of life
Normal walking velocity | 3 months
  Normal walking velocity (NW velocity, in cm/s) will also be evaluated three months after the onset of treatment as a secondary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Reto W Kressig, MD, Principal Investigator — Chair of Geriatrics, Medical Faculty, Chief, Department of Acute Geriatrics, University Hospital, Basel
Locations (1):
- Basel Mobility Center, Department of Acute Geriatrics, Basel, Switzerland

REFERENCES:
- [Derived] Hardi I, Bridenbaugh SA, Cress ME, Kressig RW. Validity of the German Version of the Continuous-Scale Physical Functional Performance 10 Test. J Aging Res. 2017;2017:9575214. doi: 10.1155/2017/9575214. Epub 2017 Jul 9. PMID 28775900